CLINICAL TRIAL: NCT04541069
Title: Enhancing Social Communication and Emotional Development in Under 5 Children: Intervention Strategies for Inclusive Child Care Practices in Bangladesh.
Brief Title: Enhancing Social Communication and Emotional Development in Under 5 Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre for Injury Prevention and Research Bangladesh (Other)
Responsible Party: Principal Investigator, Saidur Rahman Mashreky, Professor, Director, Centre for Injury Prevention and Research Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2005
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Early Childhood Developmental Disability (Disorder)

STUDY DESIGN:
Intervention Model Description: Pragmatic Cluster Randomized Trial
Who Masked: Outcomes Assessor
Masking Description: When the early childhood development assessment will be done by data collectors through ASQ insruments, they will not be aware of the respondent's status of whether they received the intervention or not.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Communication and Emotional Skill Development (SCESD) (Experimental): This arm will get the intervention which is the Early Childhood Development (ECD) training.
  Interventions: Behavioral: Social Communication and Emotional Skill Development (SCESD) module
- Control (No Intervention): This arm will not get any intervention.

INTERVENTIONS:
Behavioral: Social Communication and Emotional Skill Development (SCESD) module — The intervention, Social Communication and Emotional Skill Development (SCESD) module, is based on the basics of the neuroscience of child development. The module has focused on these basic behaviors of infants, and has incorporated strategies to enhance the five basic behaviors i.e. eye contact, attention to others, joint attention, imitation and non-verbal communication.
  Arms: Social Communication and Emotional Skill Development (SCESD)

SUMMARY:
In the United Nation's Sustainable Development Goals (SDGs), the conversation has shifted from the complexity of ensuring decrease in infant mortality to that of holistic wellbeing of children from conception onwards by ensuring early learning opportunities along with nutrition, security and safety. About 13 - 23 percent children in Bangladesh present symptoms of diagnosable and preventable mental health conditions in early childhood. The aim of this effectiveness-implementation hybrid type 2 cluster randomized trial is to implement training program to enhance parental understanding of child's social communication and emotional development, ways to support positive behavior management skills, and to enhance parents' cognizance about when professional help may be sought. Shuchona Foundation's module-based training manual on Social Communication and Emotional Skill Development (SCESD) is designed to sensitize and educate parents/ caregivers on child development. This module will be implemented in Sonargaon, Gojaria and Raiganj Upazilas. The administrative wards in the unions will serve as clusters for the study's first phase. The first phase of six months duration will explore qualitatively the adaptability of existing health system, train field level health workers, training of the data collectors on administering Ages and Stages Questionnaire (ASQ), enrol mothers for equipping them with knowledge and skill to stimulate Early Childhood Development (ECD) and identify delayed childhood development, followed by assessment of ability of mothers to note secondary outcomes or delay at the earliest. The sessions for mother will be conducted using the existing health system of Bangladesh.

A mixed-methods approach comprising of process mapping, qualitative and quantitative data analyses will be used to assess implementation of the intervention with focus on identifying failures in implementation, why they exist and how to reduce them for future implementation and scale-up.

DETAILED DESCRIPTION:
2. Introduction The last five years have witnessed a plethora of literature on early childhood development, the first 1000 days in infancy, and holistic wellbeing of children from conception onwards. In large part due to the United Nation's Sustainable Development Goals (SDGs), the conversation has shifted from the complexity of ensuring decrease in infant mortality to that of ensuring nutrition, prenatal health care, security and safety, early learning opportunities all of which work together to lead to better outcomes for children. This is a significant shift for most low and middle income countries (LMIC's), like Bangladesh, where a well-prepared plan to implement effective programs that are also low-cost and applicable to the existing infrastructure does not exist. According to the Early Childhood Nurturing Care Framework, nutrition, health, early learning, responsive caregiving, security and safety are important components that ensure that countries can achieve their SDG's and thereby enable better outcomes in later childhood and adulthood. 1 In addition, planning for an approach that ensures children at risk for conditions like autism and other developmental disorders are identified sufficiently early in infancy is an added challenge. According to Munir et al (2018), parents in LMIC's rarely reach out to health professionals for behavioral and developmental concerns due to social stigma and lack of evidence-based services, unless their child is experiencing acute medical distress. This in large part explains why, in a country like Bangladesh, which has a comprehensive policy for children, disabilities, health care and nutrition, there still continues to be delay in providing early intervention services and medical services to children with neurodevelopmental disorders.

Figure 1 The nurturing care framework (Wertlieb, 2019) Nurturing care refers to giving children the opportunity to learn in their early childhood years through interactions with peers and adults in a responsive and emotionally supportive environment, which is the result of public policies, programs, and services that include health, nutrition and security. Global research indicates that nearly 385 million children are living in extreme poverty, 155 million children under five have stunted growth, and more than 240 million affected by conflict.2-4 About 300 million children between ages two and four are regularly subjected to violent discipline, including physical punishment and psychological aggression.4 Moreover, around 250 million children (43%) less than 5 years of age in low- and middle-income countries are at risk of not reaching their developmental potential.5 Researches with 0-5-years old indicate that health risks before 24 months impacts mental development of the child. More than 200 million children under 5 years of age are not reaching their developmental potential because of poor health, lack of nutrition and poverty. Medical issues such as delivery by unskilled attendant; infections like malaria and cholera, inadequate nutrition, and inadequate stimulation significantly increase risk for disabilities and reduce the potentiality for greater success in life.6-8 Bangladesh has implemented several programs in order to mitigate the effects of poverty, prenatal and early childhood malnutrition and adverse living conditions. Programs to educate pregnant women, provide health education in communities, adequate vaccinations, stipends and various forms of nutritional programs are currently being provided in many parts of the country through a variety of programs. Nevertheless, according to the recommendations of research in the area of early childhood intervention (EDI) and inclusive early childhood education (IEDE), the most effective programs should encompass both health, learning and stimulation9,10. According to results from the INTERGROWTH-21ST Project, when adequate nutrition and education are given to primary caregivers (mostly mothers) of under two years old children, it accounts for 10% variance in the acquisition of all developmental milestones across all domains, nullifying the supposed effects of cultural child-rearing practices11.

The influence of risk and protective factors cannot be evaluated separately from each other; the balance between the burden experienced by parents, and the capacity and resources of the parents should always be evaluated together.12 A population based study in Bangladesh indicated that 14.6% of children have a diagnosable behavioral impairment13 with a higher prevalence (40.4%) among orphan children.14 Male children were found to be present with increased risk factors.15 A systematic review published in 2014 in Bangladesh indicated that 13.4 to 22.9% children in Bangladesh present symptoms of diagnosable mental health condition.16 Bronfenbrenner17 evidenced that environmental factors play a critical role in coordinating the timing and pattern of gene expression, which in turn determine initial brain architecture. He stated that the development of children is rooted within a bigger context, which includes the characteristics of both the parents and the child, and are a result of constant interaction, as one influences the other: the bioecological model of specific experiences facilitates or inhibit neuronal connectivity at key developmental stages. Our perceptual, cognitive, and emotional capabilities are built upon the platform provided by early life experiences18 It has been evidenced that knowledgeable and skilled parenting can facilitate a supportive relationship and enhance the future positive psychosocial development of the child.12

In the absence of clinically validated biomarkers and the significant variation in the presentation of milder autism cases (typically referred by clinicians as 'high functioning' autism), it is extremely necessary to find a methodology for early detection of risk factors that are easily noticeable by caregivers, coupled with intervention techniques that can be used effectively in the natural environment of the child. The median age of autism diagnosis and intervention in the United States, where tremendous awareness activities are being done, is still at 4.5 years of age. A recent review of the research on when and how parents should be informed about their child's autism diagnosis (See Figure 2) shows that although core areas of deficit in social communication and repetitive stereotypical behaviors do not become apparent till nearly 24 months of age, many early indicators do exist that have been substantiated as prodromal features in the first 6 months 20. And given our understanding of brain plasticity and developmental peaks, there is a strong likelihood that well-trained caregivers can effectively prevent core symptoms of autism from manifesting. At the very least, methods, as prescribed by the Social Communication and Emotional Skill Development (SCESD) manual, could enable a reduced intensity of the delays.

Early identification of developmental disorders is critical to the well-being of children and their families.21 The earlier identification of delay increases the opportunity to provide early intervention, maximizing the benefit of that intervention.22 Thus promoting the development of the child in later years.12 Although evidence shows that early intervention can reduce the impact on the functioning of the child and the family, identification of inadequate social communication and emotional skills in young children has always been a challenging process.22 Family members can play a vital role in the identification and application of the intervention process especially in children under 5 years of age.23 In developing countries with increased child survival, the number of children with social-communication delay is also increasing24. Convention on the Rights of the Child (CRC) and the Convention on the Rights of People with Disabilities (CRPD), both state that children with disabilities have the right to develop to their maximum potential. Investment in Early Childhood Development (ECD), should also focus on children at risk of developmental delays or disabilities24. In a report of the project "Developing an Inclusive Education and ECD Strategy" (2013-2014), Plan Sri Lanka in collaboration with the faculty of medicine university of Kelaniya recommended each early learning activity to be broken down into small steps to support children with delays/ disabilities. It also recommended that the staff/ teachers involved in pre-school cares should be well equipped with the knowledge of screening of early delays/ disabilities.

Due to lack of proper tools and resources, many children with developmental delays are not being identified early in LMICs. Moreover, after the first concern, it requires a long time to get professional help. As a result, these children often must wait until they start going to school before they receive help25. Therefore, ECD programs beside providing child development strategies also need to make parents/ caregivers aware of the stages of regular child development which will potentially enable the families to pick up any difference from the typical developmental trajectory. This will in turn help early detection of developmental delays. With proper support, these delays can be prevented from growing into a disability or reducing the severity of the disability and thereby potentially leading to lesser poverty and marginalization.

It should be noted that for LMIC's like Bangladesh, an early intervention model is needed that can be implemented by non-experts with minimal training, and at a low cost. It is also important that the model can be easily scaled up and implemented within the existing childcare service settings 26. In order to achieve these goals, Shuchona Foundation developed a training program that can be learned/adopted by parents, caregivers, daycare workers and others. The primary philosophy of the training is based on principals of the Early Start Denver Model and is focused on teaching social communication skills and behavior management techniques, which could be used within day-to-day typical childcare practices such as feeding, bathing, etc. Additionally, the current project would explore the possibility of parental skills training; in addition to a home-based early intervention model could be effectively incorporated into a variety of existing government programs.

Shuchona Foundation's module-based training manual on Social Communication and Emotional Skill Development (SCESD) is designed to sensitize and educate parents and other caregivers on the development of the child under their care. Developed in Bangladesh and field-tested, the manual is based on the premises of social interaction challenges often experienced by children with autism spectrum disorders (ASD). It is based on the premise that enabling parents to recognize early indicators of social-communication delay and teaching them simple adaptations to everyday childcare practices, may serve as an effective prevention practice that possibly could mitigate the need for further screening and/or seeking specialist care for the milder delays 27. In addition, by teaching functional strategies applicable in the natural home environment, parents with children who later receive a diagnosis and require professional intervention would find it relatively easier to implement the professional's recommendations in the home. Thus, enabling the intervention to be more effective and increasing the likelihood that the parents would be partners in the treatment process of their child over the years. Recent studies on early autism interventions indicate programs that include parent skill-building programs are a key component to ensuring that the effects of the intervention remain in later childhood and those children do better in social interactions with peers28, although existing community-based programs appear not to be as effective as those implemented in clinical settings 29. The aim of this training is to enhance parental understanding of typical child development with significant focus on social communication and emotional development; to teach parents positive behavior management skills; teach parents and other caregivers simplified evidence-based strategies that can be implemented in the typical care of their child; to enable parents to be more cognizant for when professional help needs to be sought, and be effective partners with the professionals involved in the therapeutic treatment of their child.

3. Objectives

3.1 General objective To design of a social communication and emotional skill development intervention and determine its' efficacy in promoting Early Childhood Development (ECD) and controlling developmental delay among under 5 children using existing health system in Bangladesh.

3.2 Specific objectives

1. To design and strategize a social communication and emotional skill development intervention for infants and young children in community health care settings
2. To assess the effectiveness of the community centered module-based approach in monitoring social communication and emotional development and those factors which may influence social-emotional development, in infants and young children.
3. To conduct qualitative and quantitative assessment of fidelity of the trainer pool and carers who completed the training and competency test
4. To compare the capacity/skill/competency to identify socioemotional problems among study population of trained carers to carers as usual.
5. To evaluate the predictive values of community-based approach, in accurately identifying specific social-emotional problems among sample population
6. To evaluate the quality of care and carers' compliance regarding responsive parenting, disclose concerns, as compared to carers as usual.
7. To measure sociodemographic, reproductive and anthropometric characteristics and other potential confounders of the study population
8. To use, adopt and or validate culturally sensitive, socially acceptable and scientifically rigorous research instrument for measuring the key variables of the study
9. To assess the compatibility/system/adaptability/readiness of the existing primary health care settings to integrate and deliver the proposed intervention
10. To determine the cost effectiveness of the intervention

5. Brief description of the module for intervention The intervention, Social Communication and Emotional Skill Development (SCESD) module, is based on the basics of the neuroscience of child development. Some basic behaviors in early childhood, starting from infancy can predict future cognition, socialization and language acquisition. The module has focused on these basic behaviors of infants, and has incorporated strategies to enhance the five basic behaviors i.e. eye contact, attention to others, joint attention, imitation and non-verbal communication. The development of typical brain functioning requires input via all of the major sensory systems. Therefore, different fun activities have been shown to encourage children's tactile, auditory and visual sensation.

The techniques used in this training can be used throughout the day during caregiving and other daily activities, based on the principles of the Early Start Denver Model (ESDM). ESDM, which is mainly used for children with ASD, is based on normal child development model, therefore the basic developmental stages and strategies to enhance child development in different domains can be applicable for all children. This has made the ECD module inclusive for all children and has reduced the gap between research and practice.

The module has been developed after analysing the financial and other resource support system operating in the community, and as such has incorporated evidence based measures in ESDM for encouraging parent-child dyadic interaction.

There are some chapters in the module that focus on children's 'Receptive' and 'Expressive' language development. Using non-verbal communication has also been encouraged through 'Least to Most technique'. After each chapter different stages of development on the specific topic have been described in an easy to understand way (including pictorial) to help the caregivers understand the level of functioning of the child and what steps need to be taken to advance the development. The basics of Applied Behavior Analysis (ABA) and Positive behavior Support (PSP) techniques have been explained in a way that can be translated into the real-life situation by parents and other caregivers. Two separate sections have been incorporated to encourage to support children's behaviors in a positive way. The need for setting up rules and how to do that has been explained in one. Strategies to tackle children's difficult behaviors has been discussed in another section. Besides teaching the behavioral strategies, the main focus of these chapters is to make sure that the children know about their emotions, and how to support them to express it properly; this is mainly based on the principles of children version of 'Cognitive Behavior Therapy' model. The chapter on children's attention skills and motor development has also been incorporated in the module.

There is also a small booklet for the mothers with the key messages and relevant pictorial contents. The complete module takes a total of 19 hours to be delivered. The total content is split into 4 sessions. However, for the first phase of the project, only the first 3 sessions will be provided to the mothers. These 3 sessions will be distributed between 2 classes. The first class will be 30 minutes long, the second class which will also include some activity will be an hour long. The sessions will be taken in spaced intervals, and will be delivered personally to mothers and families at households by multi-purpose volunteers.

The module was reviewed by international experts in the field of child development. Further revisions were done based on the experience and feedback from trainings conducted with different audience, including audience with limited or no literacy. The module was finalized by Shuchona Foundation Expert Team.

6. Study Overview 6.1 Study setting The study setting for this effectiveness-implementation hybrid type 2 cluster randomized trial will be in three Upazilas of Bangladesh, namely Sonargaon, Gojaria and Raiganj. Each Upazilla usually comprises of 10 unions and each union has 9 wards in it. The wards in the unions will serve as clusters for the study. Usually, there is one Upazila Health complex (UHC) in each Upazila, while each ward consists of one community clinic, and five multipurpose volunteers. The community clinics are under the supervision of respective UHC. The community clinics and Upazila Health Complexes are the primary level of health care services.

6.2 Study duration

For effective intervention, the study has been divided into four phases as shown in figure 4. The first, second, third and fourth phase will be the focus of this study which will last for about 6 months. It would be pertinent to explain the phases to highlight the content of the four phases. The first phase will include an exploration to assess whether the health system is adaptive and ready for the implementation of this project. In the second phase, training of the primary health care providers who will give antenatal services and enrolment of mothers in the study, training of the Health Assistants (HA), Family Welfare Assistant (FWA) and Community Health Care Providers (CHCP) who will work in the community at household level to deliver the training to mothers and families, and also training of the data collectors who will measure the study outcomes at household level. Second phase will start enrolling mothers of children under 2 months of age, which will continue in subsequent phases of the study. In the third phase, mothers will be trained and data will be collected on the information of child development. The later phase of the study will assess children and mothers at different stages of the children's lives.

The initial two months of the first phase will be used for qualitative data collection and, analysis, followed by designing the intervention incorporating the findings. Accordingly, antenatal care (ANC) providers, Health Assistants (HA), Family Welfare Assistant (FWA), Community Health Care Providers (CHCP), and data collectors will be trained, and enrolment of study participants will commence. During the next four months the designed intervention will be implemented, along with continuation of the enrolment of study participants. When mothers enrolled for the study have finished undergoing the training sessions, the respective children will be primarily assessed with the Ages and Stages Questionnaire (ASQ), followed by assessment of ability of mothers to note secondary outcomes or delay at the earliest.

7. Study participants 7.1 Sample and sample size calculation All available clusters (wards) will be listed in the study area and thus a sampling frame will be generated. Required number of clusters calculated during sample size estimation will be selected from this frame randomly for entering the study using a random sequence generator in Microsoft Excel. Randomization of the available clusters into intervention and control groups will be done in the same manner using random numbers. Control and intervention groups will be selected in 1:1 ratio.

All mothers (primary caregivers) of children under 2 months of age in the study area will be approached for enrolment. The calculation of sample size is as follows. Prevalence of behavior problem of young children in Bangladesh was considered as the indicator for calculating the sample size of this study. The sample size has been calculated considering the prevalence to be 14.6%.16 To measure a 35% effect size, an equal and minimum number of 624 mothers for each of the interventions and control arm will be recruited to gain a power of 80% at a 5% level of significance (two sided) with the formula for Randomized control trials. To address the cluster effect of the design, the sample size is multiplied by 1 + (m - 1)ρ, where m is the average cluster size and ρ is the is the inter cluster correlation coefficient (ICC).21,22 Considering inter cluster correlation of 0.05,22 and an average number of 10 eligible mother in each cluster the design effect is 1.45 [1+(10-1)*0.05]. Thus, we determined that we need a minimum of 905 eligible participants per arm. Considering 10% drop out the size will be 1002. Which in turn makes 101 clusters per arm. Total 2004 mother will be recruited for intervention and control arm.

7.2 Participants Recruitment The study will focus on the rural population as majority of the country's population reside in rural areas, and are less likely to be exposed to ECD interventions. Primarily, the mothers of children under 2 months of age will be continuously enrolled as study participants. These mothers will be equipped with the knowledge and skill for stimulating ECD and identifying indicators of delayed development of children (training sessions), which will take place during the Inter personal communication (IPC), and Expanded Programme on Immunization (EPI) sessions where the mothers visit to get their children vaccinated. For the first phase, data of mothers who will undergo at least 2 training sessions will only be included for analysis. The mothers will then be followed up for the next two years covering both phases. In this second phase the mother child unit who were trained will be followed every two months, as well as the enrolment and training of new mothers will continue. The family of the mother will also receive the intervention which is thought to enable a supportive environment for the mother and also due to the fact that, children are exposed to and influenced by other family members as well. Mothers, however, are the main recipient of the intervention.

The mothers will be identified at the primary health care center where they receive their antenatal check-ups. Assistance of field health workers will also be taken to identify and enroll the mothers. The health care provider at the center or field health workers will be responsible for taking consent, recording the enrolment of the eligible participant in the intervention and control clusters, and taking anthropometric measurements of all enrolled mothers. After randomization, the mothers enrolled in the control clusters of this study will receive conventional antenatal care. The contact information of these mothers will be collected and maintained by the manager of the primary health care center where mother receives antenatal service. This information will then be passed on to the Coordinators who will then coordinate with the data collectors.

Inclusion Criteria:

* Mother of children under 2 months of age
* Eligible mother who will give consent to participate in the study

Exclusion Criteria:

* Mothers with a critical illness that prevents them to take part in the training sessions or to take care of the child
* Families that intend to move out of the area within the study period

7.3 Intervention distribution

Distribution of Upazillas, Unions, and wards:

1. There are 3 Upazillas (Nandail, Savar and Raiganj)
2. Total 33 Unions (13 Unions in Nandail, 12 Unions in Savar, and 9 Unions in Raiganj).
3. We will take about 9 to 10 Unions from each Upazilla
4. So total 27 to 30 Unions
5. Total about 297 wards. We will take 243 to 270 wards
6. According to sample size calculation we need 202 wards (clusters) randomly selected from these 243 to 270.
7. 101 of the wards will be randomly assigned to intervention arm and another 101 wards will be randomly assigned to control arm
8. Total of 7 wards per Union will be selected.
9. 3-4 intervention ward per Union and 3-4 control ward per Union

Who will be assigned work at each level

1. Each Union will have a Union supervisor
2. So 27 to 30 Union Supervisors
3. Each ward has a health assistant (HA) under it
4. There will be one multipurpose volunteer per Union Role of individuals at each level

1. Union supervisors:

* Make sure that the mothers are informed about the trainings
* Make sure that trainings are carried out at EPI session nearest to the enrolled/identified mothers
* Make sure that the mothers go to that EPI session and gets the SCESD training session
* Will know the exact age of the child
* Will schedule the points of data collection for each of the child accordingly (at 2 months, 6 months, 12 months, and 18 months)
* Will keep track of the number of training sessions received by each of the mother
* This tracking has to be done for about 36 mother-child pair for each Union supervisor at each Union 2. Health assistants (HA):
* Deliver the training sessions every month according to schedule
* Training sessions concurrently with the EPI sessions as per necessity
* Total of 9-12 mother-child pair at each ward will receive the training sessions.
* Help in identifying and enrolling mothers for intervention (See "Enrollment of mothers) 3. Multipurpose Volunteers (MPV):
* Deliver training sessions every month when a mother who is enrolled misses a session at the EPI
* Follow schedule for the training to individual mother
* Make sure total of 9 to 12 mothers receive the SCESD training per ward
* Help in identifying and enrolling mothers for intervention (See "Enrollment of mothers)

7.4 Guidelines for field work during COVID-19 Purpose of the Guideline This guideline will provide direction and outline social interaction during the COVID-19 pandemic situation. The focus of this document is maintaining proper social distancing and protective measurements that will ensure to reduce the negative impact on health and social impacts.

ELIGIBILITY:
Inclusion Criteria:

* Mother of children under 2 months of age
* Eligible mother who will give consent to participate in the study

Exclusion Criteria:

* • Mothers with a critical illness that prevents them to take part in the training sessions or to take care of the child

  * Families that intend to move out of the area within the study period

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2004 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
ASQ score (Ages and stages questionnaire) score | 6 months
  To assess the effectiveness of the community centered module-based approach in monitoring social communication and emotional development and those factors which may influence social-emotional development, in infants and young children, this instrument will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Saidur R Mashreky, Phd, Principal Investigator — Director